CLINICAL TRIAL: NCT03297255
Title: Factors Influencing the Occurrence and Long-term Survival of Patients With Primary Liver Cancer: A Cohort Study in South China
Brief Title: Primary Liver Cancer Cohort of South China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: SYS-2013
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Primary Liver Cancer
Keywords: Primary Liver Cancer; Cohort Study
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and liver tissue were retented during therapy

SUMMARY:
This longitudinal observational cohort study was designed to investigate factors that influencing the occurrence and long-term survival of patients with primary liver cancer. Basic informations and detailed diagnosis informations (AJCC/TNM stage, MELD score, Child-Pugh score, and BCLC stage) were collected by professional doctors. Clinical outcomes (death, recurrence, and metastasis) will be followed up every two years after therapy.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is highly malignant with high mortality which is particularly popular in China. Many factors are believed to associate with the occurrence and prognosis of liver cancer. This longitudinal observational cohort study was designed to investigate factors that influencing the occurrence and long-term survival of patients with primary liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* consistent with primary liver cancer diagnostic criteria
* first diagnosis (from diagnosis to admission interval of less than a month)
* did not do any treatment of liver cancer

Exclusion Criteria:

* refused to participate in this study
* suffering from more than two kinds of primary tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of this study were invited from Sun Yat-sen University Cancer Center as soon as they were diagnosed as primary liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time of Death | Up to 10 years
  The exact death time of each participants will be checked in the government medical records system

SECONDARY OUTCOMES:
Time of recurrence | From date of diagnosis until the date of cancer recurrence or date of death from any cause, whichever came first, assessed up to 10 years
  Time of recurrence will be obtained by telephone interview or medical treatment records
Time of metastasis | From date of diagnosis until the date of cancer metastasis or date of death from any cause, whichever came first, assessed up to 10 years
  Time of metastasis will be obtained by telephone interview or medical treatment records

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Huilian, Professor, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu ZY, Yishake D, Fang AP, Zhang DM, Liao GC, Tan XY, Zhang YJ, Zhu HL. Serum choline is associated with hepatocellular carcinoma survival: a prospective cohort study. Nutr Metab (Lond). 2020 Mar 30;17:25. doi: 10.1186/s12986-020-00445-z. eCollection 2020. PMID 32256673
- [Derived] Liu ZY, Tan XY, Li QJ, Liao GC, Fang AP, Zhang DM, Chen PY, Wang XY, Luo Y, Long JA, Zhong RH, Zhu HL. Trimethylamine N-oxide, a gut microbiota-dependent metabolite of choline, is positively associated with the risk of primary liver cancer: a case-control study. Nutr Metab (Lond). 2018 Nov 20;15:81. doi: 10.1186/s12986-018-0319-2. eCollection 2018. PMID 30479648